CLINICAL TRIAL: NCT01753271
Title: Subacute Effects of Cervicothoracic Spinal Manipulation in Addition to Shoulder Manual Therapy Plus Exercise Intervention in Individuals With Subacromial Impingement Syndrome: a Randomized, Controlled Clinical Trial Pilot Study
Brief Title: Subacute Effects of Spinal Mobilization to Treat Subacromial Impingement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: High Point University (Other)
Collaborators: University of Illinois at Chicago (Other); Walsh University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201208-122
Record Dates: First submitted 2012-12-11; First posted 2012-12-20 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Subacromial Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thoracic Mobilization (Experimental): thoracic mobilization in addition to shoulder mobilization plus exercise
  Interventions: Other: thoracic mobilization & shoulder mobilization & exercise; Other: shoulder mobilization & exercise
- exercise only (Active Comparator): shoulder mobilization plus exercise alone
  Interventions: Other: shoulder mobilization & exercise

INTERVENTIONS:
Other: thoracic mobilization & shoulder mobilization & exercise
  Arms: Thoracic Mobilization
Other: shoulder mobilization & exercise

SUMMARY:
Specific Aims and Hypotheses Aims To investigate the incremental benefits of cervicothoracic spinal manipulation in addition to shoulder mobilization and exercise for improving range of motion, pain, physical function and fear avoidance beliefs in patients with subacromial shoulder impingement.

Hypotheses It is hypothesized that those subjects who receive spinal manipulation in addition to shoulder mobilization and exercise will achieve greater improvements in range of motion, pain, function and fear avoidance beliefs at two weeks following treatment conclusion, at 4 weeks following treatment conclusion, and at discharge when compared to the subjects who did not receive the spinal manipulation.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible, participants must meet the clinical prediction rule for unilateral subacromial shoulder impingement including: a) positive Hawkins-Kennedy impingement sign, b) positive painful arc sign, and c) weakness in external rotation with the arm at the side

Exclusion Criteria:

* Individuals with contraindications to treatment with mobilization and manipulation (Appendix A) will be excluded

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index Change over time | 2 weeks, 4 weeks, discharge
  Patients will be followed for the duration of their physical therapy treatment. An average of 12 visits over 6 weeks

SECONDARY OUTCOMES:
Numeric Pain Rating Scale change over time | 2 weeks, 4 weeks, discharge
  Patients will be followed for the duration of their physical therapy treatment. An average of 12 visits over 6 weeks
Fear Avoidance Beliefs Questionnaire change over time | 2 weeks, 4 weeks, discharge
  Patients will be followed for the duration of their physical therapy treatment. An average of 12 visits over 6 weeks

OTHER OUTCOMES:
Shoulder range of motion change over time | 2 weeks, 4 weeks, discharge
  Patients will be followed for the duration of their physical therapy treatment. An average of 12 visits over 6 weeks
test of resistance change over time - number of repetitions performed | 2 weeks, 4 weeks, discharge
  The test is performed by asking the patient to hold the shoulder at 90 degrees of shoulder flexion and follow a 20cm wide spiral using their affected arm. The patient is asked to complete as many spiral movements as possible until stopped secondary to pain. The maximum number of repetitions to be performed is 20.
  Patients will be followed for the duration of their physical therapy treatment. An average of 12 visits over 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alexis A Wright, Phd, Principal Investigator — High Point University
Locations (3):
- United States (3):
  - University of Illinois at Chicago, Chicago, Illinois
  - Physical Therapy Services, Elizabethton, Tennessee
  - East Tennessee State University, Johnson City, Tennessee

REFERENCES:
- [Derived] Wright AA, Donaldson M, Wassinger CA, Emerson-Kavchak AJ. Subacute effects of cervicothoracic spinal thrust/non-thrust in addition to shoulder manual therapy plus exercise intervention in individuals with subacromial impingement syndrome: a prospective, randomized controlled clinical trial pilot study. J Man Manip Ther. 2017 Sep;25(4):190-200. doi: 10.1080/10669817.2016.1251377. Epub 2016 Nov 7. PMID 28912631